CLINICAL TRIAL: NCT00003461
Title: Phase I Study of At-Labeled Anti-Tenascin Human/Mouse Chimeric Monoclonal Antibody 81C6 (ch81C6) Via Surgically Created Cystic Resection Cavity in the Treatment of Patients With Primary or Metastatic Brain Tumors
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Primary or Metastatic Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 2237; DUMC-2237-01-12R4; DUMC-0013-00-1R2; DUMC-0036-99-1R1; DUMC-060-98-1; DUMC-2237-00-12R3; DUMC-98007; NCI-5P50NS20023; NCI-G98-1462; CDR0000066493
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer; Neuroblastoma
Keywords: localized resectable neuroblastoma; recurrent neuroblastoma; recurrent adult brain tumor; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; adult oligodendroglioma; tumors metastatic to brain; adult anaplastic astrocytoma; adult mixed glioma; adult pineal parenchymal tumor; adult central nervous system germ cell tumor; adult grade III meningioma; adult pilocytic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Neuroblastoma; Brain Neoplasms; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Oligodendroglioma; Astrocytoma; Glioma; Pinealoma; Gliosarcoma | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Procedure: surgical procedure
Radiation: astatine At 211 monoclonal antibody 81C6

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver radioactive tumor-killing substances to them without harming normal cells. This may be effective treatment for primary or metastatic brain tumors.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy in treating patients with primary or metastatic brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of monoclonal antibody (MAb) Astatine At 211 Antitenascin Human/Mouse Chimeric 81C6 (At 211 MAb 81C6) therapy delivered via the intracranial resection cavity in patients with recurrent primary or metastatic malignant brain tumors.
* Identify objective therapeutic responses of these patients to this treatment.

OUTLINE: This is a dose escalation study.

Patients undergo surgical resection of their tumor at which time an indwelling intracranial resection cavity catheter is surgically placed. Patients receive one dose of astatine At 211 antitenascin monoclonal antibody 81C6 (At 211 MAb 81C6) via the intralesional catheter.

Cohorts of 3-6 patients are treated at escalating doses of At 211 MAb 81C6. The maximum tolerated dose is the highest dose at which no more than 3 of 6 patients experience dose limiting toxicity.

Patients are followed initially at 4 weeks, then at approximately 12 weeks, at 24 weeks, and then every 12 weeks for 1 year.

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed or recurrent supratentorial primary or metastatic malignant brain tumor
* Measurable disease by MRI or CT scan

  * Candidate for surgical resection
  * Extension of tumor no more than 1.0 cm beyond the margin of the surgical cavity
* Demonstrated reactivity of tumor cells with tenascin by immunohistology with either a polyclonal rabbit antibody or the monoclonal mouse antibody
* No infratentorial tumors, diffusely infiltrating tumors, tumors with subependymal spread, or multifocal tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Alkaline phosphatase less than 1.5 times normal
* SGOT less than 1.5 times normal

Renal:

* Creatinine less than 1.2 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 weeks since prior chemotherapy, unless unequivocal evidence of progression

Endocrine therapy:

* Concurrent corticosteroids allowed, but must be on stable dose for at least 1 week

Radiotherapy:

* At least 3 months since prior radiotherapy to site of measurable disease in the CNS

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States